CLINICAL TRIAL: NCT05707702
Title: Lactobacillus Lozenges as Preventative Care in Low-grade Dysplasia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study did not start as a key co-investigator left the institution.
Sponsor: Boston Medical Center (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-42906
Record Dates: First submitted 2022-12-10; First posted 2023-02-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Low-grade Oral Dysplasia
Keywords: Probiotic lozenge; Oral cavity squamous cell carcinoma; Oral microbiome
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic lozenges (Experimental): Participants in this arm will be be instructed to take a lozenge daily for 6 weeks. They will also receive oral dysplasia standard of care.
  Interventions: Biological: Probiotic oral lozenges
- Standard of care for oral dysplasia (Active Comparator): Participants in this arm will receive oral dysplasia standard of care.
  Interventions: Other: Standard of care for oral dysplasia

INTERVENTIONS:
Biological: Probiotic oral lozenges — Participants in this arm will be be instructed to take a lozenge daily for 6 weeks. They will also receive oral dysplasia standard of care.
  Other Names: FLORASSIST® Oral Hygiene lozenges
  Arms: Probiotic lozenges
Other: Standard of care for oral dysplasia — Oral dysplasia standard of care includes clinical surveillance and risk factor reduction (such as smoking cessation).
  Arms: Standard of care for oral dysplasia

SUMMARY:
There are limited evidence-based management options for patients with low-grade oral dysplasia. Despite the risk of malignant transformation, management is frequently limited to risk factor reduction (such as smoking cessation) and clinical surveillance. An intervention for low-grade oral dysplasia which could induce regression or decrease rates of malignant transformation has the potential to be a valuable preventative tool to reduce rates of oral cancer.

The investigators will conduct a randomized clinical trial to investigate if the administration of a probiotic lozenge to patients with low-grade oral dysplasia result in decreased peri-tumoral inflammation as evidenced by impacts on populations of tumor-associated macrophages and tumor-infiltrating lymphocytes, and decreased dysbiosis at the disease site compared with the contralateral normal site. The investigators hypothesize that these changes may increase the rate of clinical regression of these lesions.

ELIGIBILITY:
Inclusion Criteria:

* Presence of biopsy-proven low-grade or mild oral dysplasia

Exclusion Criteria:

* Active oral cavity malignancy
* Active oral cavity high grade dysplasia
* Currently undergoing chemotherapy or immunotherapy, or have used these agents within the prior 6 months
* History of external beam radiation therapy to the head and neck area
* Diagnosis of HIV with decreased CD4 count and/or detectable viral load
* Current use of systemic or orally absorbed steroids
* Patient undergoing stem cell transplantation
* Patients taking anti-rejection medication after stem cell or solid organ transplantation
* Patients using injectable immunosuppressive drugs for autoimmune disease
* Pregnant or nursing women
* Patients who are hospitalized
* Patients with a heart valve abnormalities or a history of valve replacement or endocarditis
* Patients with active severe acute intestinal disease (active bowel leak, acute abdomen, active colitis) or a history of short bowel syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04-29 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Clinical regression of dysplastic lesion | 6 weeks
  This outcome will be assessed using blinded review of clinical photographs and measurements of the lesions to determine if the lesion has regressed, remained the same or progressed since baseline.

SECONDARY OUTCOMES:
Microbiome at the lesion site | baseline, 6 weeks, 12 weeks
  The microbiome at the lesion site will be compared with the contralateral normal tissue to determine whether the dysbiotic oral microbiome will show a reduction in the abundance of oral cancer-associated microbial populations after treatment with the probiotic lozenge, and whether any changes seen will persist after cessation of treatment. The analysis of the microbiology specimens will include 16s sequencing and analysis.
Change in peri-tumoral inflammation | baseline, 6 weeks
  Peri-tumoral inflammation will be assessed by analyzing populations of tumor-associated macrophages and tumor-infiltrating lymphocytes in the biopsy performed after 6 weeks of treatment compared to the pre-treatment biopsy.
Oral dysplasia lesions at 12 weeks | 12 weeks
  This outcome will be assessed using blinded review of clinical photographs and measurements of the lesions to determine if the lesion has regressed, remained the same or progressed.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Edwards, MD, Principal Investigator — Boston Medical Center, Otolaryngology
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No